CLINICAL TRIAL: NCT04887246
Title: Monitoring the Effectiveness and Safety of Covid-19 Vaccines in the University Population-National University of Colombia
Brief Title: Monitoring the Effectiveness and Safety of COVID-19 Vaccines at National University of Colombia
Status: Completed | Type: Observational
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Other Study IDs: 52932
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Covid19; SARS-CoV2 Infection
Keywords: Covid-19; Vaccines; Safety and Effectiveness
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UNISALUD population: Refers to all affiliated members or beneficiaries of the UNISALUD entity, who got any of tthe COVID-19 vaccines available in Colombia
  Interventions: Biological: COVID-19 vaccines

INTERVENTIONS:
Biological: COVID-19 vaccines — COVID-19 vaccines available at Colombia

SUMMARY:
There are relevant questions that need to be answered about the effectiveness and safety of COVID-19 vaccines. The objective of this observational study is to follow up the clinical outcomes after vaccination in all the headquarters of the National University of Colombia. It is a project that is considered institutional importance and is part of the actions that the National University of Colombia has proposed to the national government to accompany the national vaccination program.

The proposed follow-up includes the sociodemographic, cultural, clinical and pharmacological characterization of the vaccinated population, including the report of adverse events occurring after the vaccination process, the behavior of the population after the administration of the vaccine, monitoring serological outcomes, identification of medication errors and therapeutic failure. Three stages are proposed in which the population affiliated to UNISALUD is gradually included, then the beneficiaries and later the student community and their families.

The scope of the attached protocol includes Stage I, which corresponds to teachers and administrative staff (active and retired) linked to UNISALUD.

DETAILED DESCRIPTION:
OBJECTIVE: To evaluate the clinical outcomes and adverse events associated with immunization (ESAVI) of vaccines against COVID-19 in the cohort of the university community, affiliates and beneficiaries of UNISALUD and students of the National University of Colombia.

METHODOLOGY: Descriptive longitudinal, prospective and observational study. Follow-up to a cohort without a control group. Modular multi-center stage study. The development of the research is proposed through a modular, multicenter and staged study. For the first phase, all employees of the National University of Colombia (active and retired) who agree to participate in the study will be monitored. The second phase includes monitoring the beneficiaries of UNISALUD affiliates and the third phase includes students and their families. For the calculation of the sample size in phase III, it will be carried out by applying formulas for descriptive studies.

Follow-up Time: It is estimated to be one year from the date of the first dose of the vaccine. A second phase is expected to follow up the outcomes for another additional year.

Data collection: It will begin with the presentation of the informed consent for the presentation of the study. Subsequently, a periodic follow-up will be carried out via telephone or email to identify and complete the established sociodemographic, cultural, clinical and pharmacological variables.

Serological Follow-up: The humoral immune response and its duration will be analyzed through serological tests with a blood sample to a sample of the study population. Serological follow-up will be carried out in 3 moments: prior to vaccination, after the first dose of the vaccine, and at the end of the study. The collected samples will be taken to the Laboratory of the Faculty of Medicine of the National University of Colombia for their separation. Antibody analysis will be done by chemiluminescence using the Advia Centaur COV2 platform from Siemens (3).

ETHICAL ASPECTS: This research is considered a research with minimal risk (Resolution No. 008430 of October 4, 1993 in article 11 of Colombia's Ministry of Healt ). When handling very sensitive information, the informed consent of the user and / or his manager will be filled out, prior to the start of the application of the data collection instrument, and the collection of blood samples for serological monitoring.

Access to the clinical and pharmacological information of the participants affiliated and beneficiaries of UNISALUD will be required, which will be provided by the same entity, as well as the databases adjusted to the vaccination phases in Colombia. In the case of students, basic contact information and financial situation will be needed, which will be reported by the University Welfare Directorate.

The treatment of information and data collected in accordance with Law 1266 of 2008 "Habeas Data" and subject to acceptance by the participants through informed consent.

This study protocol has the endorsement of the ethics committee of the Faculty of Sciences in a meeting held on March 1, 2021 (Minutes 02-2021).

ELIGIBILITY:
Inclusion Criteria:

* All UN contractors (administrative, teachers and pensioners) who belong to the different UN headquarters and agree to participate in the study

Exclusion Criteria:

* Contractors not not affiliated to UNISALUD

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort of the university population (UNISALUD affiliated and beneficiary personnel, students and their families),
Sampling Method: Non-Probability Sample
Enrollment: 4078 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Adverse events | One year
  Reports of Adverse Events Associated with COVID-19 Vaccines
COVID-19 diagnosis | One year
  People who after the vaccination process are diagnosed with COVID-19

SECONDARY OUTCOMES:
Serological response | One year
  Serological analysis to identify humoral immune response and duration

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Nacional de Colombia, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided